CLINICAL TRIAL: NCT04996238
Title: COVACC2: Local and General Immune Response After COVID-19 Vaccination in Volunteers
Brief Title: Local and General Immune Response After Coronavirus Disease (COVID-19) Vaccination in Volunteers
Acronym: COVACC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); Vlaams Instituut voor Biotechnologie (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BC-09476
Record Dates: First submitted 2021-07-05; First posted 2021-08-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Covid19
Keywords: serum; nasal secretions; immune response
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood and nasal fluid sampling before and after COVID-19 vaccination (Other): Blood and nasal fluid will be collected just before the first vaccination (T1: pre-vaccination), between 14 and 30 days after the second vaccination (T2: post-vaccination), 6 months after the second vaccination (T3: 6 months post-vaccination), between 14 and 30 days after the third/booster vaccination (T4: post-booster-vaccination) and 6 months after the third/booster vaccination (T5: 6 months post-booster-vaccination)
  Interventions: Procedure: Blood and nasal fluid sampling before and after COVID-19 vaccination

INTERVENTIONS:
Procedure: Blood and nasal fluid sampling before and after COVID-19 vaccination — Blood and nasal fluid sampling take place just before the first COVID-19 vaccination and at 14-30 days after the second dose with the same vaccine. Sampling will be repeated at 6 months after the second vaccination, at 14-30 days after the third vaccination and at 6 months after the third vaccination. At all moments, a questionnaire is filled in.

SUMMARY:
This study aims to gain more insight in the immunological characteristics and immune response on a local level (the nose) and systemic level (the blood) of healthy people vaccinated with the current available COVID-19 messenger ribonucleic acid (mRNA; BNT162b2) and viral vector based (ChAdOx1) vaccines.

DETAILED DESCRIPTION:
The immunological assays that will be performed on blood include immunophenotyping, serologic testing and cytokine analysis. Deep characterization of patients' immune profile offers a unique opportunity for comprehensive understanding of the mechanisms behind severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) vaccination. The investigators will study immunological functions on the level of both adaptive and innate immunity by performing extensive immunophenotyping, cytokine analysis and RNA sequencing analysis. Biomarker analysis will be performed on protein and on RNA single cell level. Infectivity of different cell types including macrophages will performed. These analyses will be performed at the Human Immunodeficiency Virus (HIV) Cure Research Center (HCRC) laboratory.

Nasal fluid: The investigators will compare the immune response and immunoglobulin production in nasal secretions before and after SARS-CoV2 vaccination. The investigators aim to compare the local versus the systemic (blood/serum) response to SARS-CoV2 vaccination. Further, patients that had a proven SARS-CoV2 infection will be compared with patients that never had COVID-19 symptoms nor antibodies.

Questionnaire: a questionnaire will be filled in by the individual to assess if the individual went through a previous SARS-CoV2 infection and experienced symptoms post vaccination. The questionnaires are available as supplementary documents.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-100 years)

Exclusion Criteria:

* People with a compromised immune system Active treatment with chemotherapy HIV infection with cluster of differentiation 4 (CD4) count below 200/µl Combined immunodeficiency Treatment with methylprednisolone >16mg for more then 2 weeks Transplant patients Diagnosed Chronic Rhinosinusitis with Nasal Polyps
* Known pregnancy at the time of screening
* Inability to give informed consent or absence of legal representative who can give informed consent.
* Any contra indication for receiving the SARS-CoV2 vaccination

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Change in SARS-CoV-2 neutralization antibody levels. | Nasal secretions and serum will be collected just before the first vaccination (T1: pre-vaccination) and between 14 and 30 days after the second vaccination (T2: post-vaccination)
  In vitro qualitative determination of SARS-CoV-2 neutralization antibody in nasal secretions and serum.

SECONDARY OUTCOMES:
Change in tumor necrosis factor alpha (TNF-α) levels. | Blood will be collected just before the first vaccination (T1: pre-vaccination) and between 14 and 30 days after the second vaccination (T2: post-vaccination)
  Quantitative measurement of TNF-α in blood using an immunoassay.
Change in interferon gamma (IFN-γ) levels. | Blood will be collected just before the first vaccination (T1: pre-vaccination) and between 14 and 30 days after the second vaccination (T2: post-vaccination)
  Quantitative measurement of IFN-γ in blood using an immunoassay.
Change in interleukin 2 (IL-2) levels. | Blood will be collected just before the first vaccination (T1: pre-vaccination) and between 14 and 30 days after the second vaccination (T2: post-vaccination)
  Quantitative measurement of IL-2 in blood using an immunoassay.
Change in interleukin 1 (IL-1) levels. | Blood will be collected just before the first vaccination (T1: pre-vaccination) and between 14 and 30 days after the second vaccination (T2: post-vaccination)
  Quantitative measurement of IL-1 in blood using an immunoassay.
Change in interleukin 18 (IL-18) levels. | Blood will be collected just before the first vaccination (T1: pre-vaccination) and between 14 and 30 days after the second vaccination (T2: post-vaccination)
  Quantitative measurement of IL-18 in blood using an immunoassay.
Change in granulocyte-macrophage colony-stimulating factor (GM-CSF) levels. | Blood will be collected just before the first vaccination (T1: pre-vaccination) and between 14 and 30 days after the second vaccination (T2: post-vaccination)
  Quantitative measurement of GM-CSF in blood using an immunoassay.
Change of subsets of T cells with markers Cluster of Differentiation 69 (CD69), CD40 ligand (CD40L), CD137. | Blood will be collected just before the first vaccination (T1: pre-vaccination) and between 14 and 30 days after the second vaccination (T2: post-vaccination)
  Quantitative measurement of subsets of COVID-19 specific T cell responses with markers of immune activation using flow cytometry.
Change of SARS-CoV-2 Spike Receptor Binding Domain (RBD) binding B cells. | Blood will be collected just before the first vaccination (T1: pre-vaccination) and between 14 and 30 days after the second vaccination (T2: post-vaccination)
  Quantitative measurement of SARS-CoV-2 Spike RBD binding B cells using flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Linos Vandekerckhove, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, East Flanders, Belgium